CLINICAL TRIAL: NCT06107309
Title: Suppressive Antibiotic Therapy for Prosthetic Valve or Implantable Device Related Infectious Endocarditis
Brief Title: Suppressive Antibiotic Therapy for Endocarditis
Acronym: SATIE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8900
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Endocarditis
Keywords: Endocarditis; Antibiotic therapy; Suppressive antibiotics; Long term treatment
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endocarditis are deadly infections, which nowadays occurs mainly among older patients with multiple comorbidities. The incidence is notably high among patients with valvular prosthetic or implantable devices. Management of such situation usually requires intravenous antibiotic therapy along with removal of the infected prosthetic or device. However, such invasive procedures and revision surgeries may be judged unreasonable among these patients, who are then exposed to a high risk of infectious relapse when curative antibiotics are discontinued.

In these situation, a long-course antibiotic therapy may be used in order to maintain lasting infection control, to limit the risks of relapse of infection due to the infected device retention, and ultimately to prolong survival. This strategy is already suggested in case of infected prosthesis joint retention (IDSA 2013), and has been proposed for implantable device retention by the American Heart Rhythm Society in 2017, but data regarding its modalities and outcomes are scare.

The objectives of this study are to describe the survival of patient under long-term antibiotic therapy for endocarditis, at 6-months and 1 year after initiation. Secondary outcomes includes modalities of the suppressive treatment prescribed, its security (secondary effects, tolerance) and to precise causes of death.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject having benefited from suppressive antibiotic therapy after collegial decision in CPR Endocarditis during the period from January 1, 2016 to January 31, 2023
* Subject not opposing the reuse of their data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Death or loss of sight of the patient before initiation of suppressive antibiotic therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) having benefited from suppressive antibiotic therapy after collegial decision in CPR Endocarditis during the period from January 1, 2016 to January 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Survival of the patient who benefited from suppressive antibiotic therapy | Survival at 6 months, 1 year, 3 years after infection

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France